CLINICAL TRIAL: NCT02574793
Title: Characteristics of Glycemic Fluctuations in Newly Diagnosed Growth Hormone-Secreting Pituitary Adenoma and Cushing Syndrome Subjects
Brief Title: Glycemic Fluctuations in Newly Diagnosed Growth Hormone-Secreting Pituitary Adenoma and Cushing Syndrome Subjects
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, xiaolong zhao, Principal Investigator, Clinical Associate Professor of Endocrinology department, Huashan Hospital
Other Study IDs: KY2015-152
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2014-12

CONDITIONS: Pituitary Adenoma
Keywords: Glucose Fluctuation; GH-Secreting Adenoma; Cushing Syndrome
MeSH Terms: conditions — Pituitary Neoplasms; Cushing Syndrome | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: continuous glucose monitoring — Patients newly diagnosed GH-releasing pituitary adenoma or Cushing Syndrome in our department will be monitored blood glucose by CGMS Gold.

SUMMARY:
Glucose fluctuations present not only in patients with diabetes mellitus but also in subjects with normal glucose tolerance or impaired glucose regulation. People with Growth Hormone-Secreting Pituitary Adenoma and Cushing Syndrome are at risk of impaired glucose metabolism. Glycemic variability is poorly studied in the nondiabetic individuals. The aim of the study is to investigate the characteristics of glucose fluctuations in the newly diagnosed Growth Hormone-Secreting Pituitary Adenoma and Cushing Syndrome individuals.

DETAILED DESCRIPTION:
Glucose fluctuations present not only in patients with diabetes mellitus but also in subjects with normal glucose tolerance or impaired glucose regulation. Compared with traditional monitoring methods, continuous glucose monitoring system(CGMS) techniques provides a much more detailed understanding of shifting blood glucose levels throughout the day.It is considered reliable to evaluate glucose variability not only in patients with diabetes but also in nondiabetic individuals.

People with Growth Hormone-Secreting Pituitary Adenoma and Cushing Syndrome are at risk of impaired glucose metabolism and developing diabetes mellitus.Some researchers have shown that 15-30% Growth Hormone-Secreting Pituitary Adenoma are suffering from diabetes, 15-36% impaired glucose regulation. The rate of Cushing Syndrome individuals is 10-30% and 40-45% separately.

Glycemic variability is poorly studied in the nondiabetic individuals and has not been studied in the newly diagnosed Growth Hormone-Secreting Pituitary Adenoma and Cushing Syndrome individuals. In this study CGM was used to dynamically monitor patients being newly diagnosed with Growth Hormone-Secreting Pituitary Adenoma and Cushing Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* •newly diagnosed GH-releasing pituitary adenoma
* •newly diagnosed Cushing Syndrome

Exclusion Criteria:

* •history of diabetes mellitus and being treated with drugs
* •being treated with drugs which affect glucose metabolism in the lately 3 months
* •with other hormones affecting glucose metabolism secreted abnormally by pituitary
* •serious comorbidity like malignant tumour, severe hepatosis or nephropathy, serious hypertension(blood pressure> 180/110mmhg)
* •pregnant or breastfeeding women
* •patients allergic to patches or metal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly diagnosed GH-releasing pituitary adenoma or Cushing Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-07 (Actual)

PRIMARY OUTCOMES:
Continuous glucose profiles of mean data of 24-hour continuous glucose monitoring by the CGMS Gold | 3 days
  The monitoring results consisted of one curve and 5 parameters

SECONDARY OUTCOMES:
The mean amplitude of glycemic excursion of newly diagnosed GH adenoma patients | 3 days
  The mean amplitude of glycemic excursion of newly diagnosed GH adenoma patients during the 3 days monitored by CGMS Gold
The mean amplitude of glycemic excursion of newly diagnosed Cushing Syndrome patients during the 3 days monitored by CGMS Gold | 3 days
  The mean amplitude of glycemic excursion of newly diagnosed Cushing Syndrome patients during the 3 days monitored by CGMS Gold
The correlation of MAGE and IGF-1 in newly diagnosed GH adenoma patients | 6 months
  By compared with the outcomes after treated by SSAs or surgery we want to get weather there is a correlation between MAGE and IGF-1 in GH adenoma patients
The correlation of MAGE and cortison in newly diagnosed Cushing Syndrome patients | 6 months
  By compared with the outcomes after treated by surgery we want to get weather there is a correlation between MAGE and cortison in Cushing Syndrome patients

CONTACTS AND LOCATIONS:
Overall Officials: yiming li, Study Director — director of the endocrinology department
Locations (1):
- Xiaolong Zhao, Jing’an, Shanghai Municipality, China